CLINICAL TRIAL: NCT00499096
Title: Cardiovascular Risk Factors in Veterans With Bipolar Disorder
Brief Title: Self-Management Addressing Heart Disease Risk Trial
Acronym: SMAHRT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: MHBA-018-06F
Record Dates: First submitted 2007-07-09; First posted 2007-07-11 (Estimated); Results first posted 2014-11-20 (Estimated); Last update posted 2014-11-20 (Estimated); Status verified 2014-11

CONDITIONS: Bipolar Disorder; Cardiovascular Disease
Keywords: Chronic Illness; Disease management; Health Behaviors; Mood Disorders-Bipolar
MeSH Terms: conditions — Bipolar Disorder; Cardiovascular Diseases; Chronic Disease; Health Behavior | interventions — Chronic Care Model; MD1

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Chronic Care Model for Bipolar Disorder (Experimental): An intervention group of patients with bipolar disorder and 1 or more risk factor for cardiovascular disease; group will receive self-management group sessions, followed by phone contacts by the Care Manager. This is the chronic care model for bipolar disorder
  Interventions: Behavioral: Chronic care model for Bipolar Disorder
- Enhanced Usual Care (No Intervention): A group of patients with bipolar disorder and one or more risk factors for cardiovascular disease will be randomized to receive enhanced usual care. This group will receive usual care, plus mailings on wellness topics (attention control), and their providers will receive information on guideline concordant care.

INTERVENTIONS:
Behavioral: Chronic care model for Bipolar Disorder — The behavioral intervention is based on the Chronic Care Model (CCM) where patients receive information on managing bipolar symptoms and health habits in a group self-management session (up to 6 weekly sessions). The Care Manager then follows up with patients via phone contacts for 12 months following the intervention. The providers receive information on guidelines for care.
  Arms: Chronic Care Model for Bipolar Disorder

SUMMARY:
The purpose of this research study is to learn whether or not people with bipolar disorder can reduce their risk of heart disease and related conditions by having a Care Manager provide self management and care management.

DETAILED DESCRIPTION:
Background: Bipolar disorder is associated with significant personal and societal costs, and represents a substantial burden to the VA. Medical conditions, notably cardiovascular disease (CVD), are substantial contributors to increased morbidity and mortality in patients with bipolar disorder, in part because of behavioral and treatment factors. Despite the existence of effective medications for managing CVD-related risk factors (e.g., hypertension, hyperlipidemia, diabetes, obesity), outcomes for these conditions remain suboptimal among patients with bipolar disorder.

Objectives: The immediate objective of this study is to determine whether a manual-based Chronic Care Model (CCM) intervention compared to usual VA care improves control of intermediate physiological measures that represent risk factors of CVD for veterans with bipolar disorder. We hypothesize that, within 12 months of the intervention initiation, patients receiving the CCM intervention will be more likely to demonstrate improved control of CVD-related risk factors (blood pressure, fasting cholesterol) and report improved physical health-related quality of life.

Methods: This is a prospective, randomized, controlled, single-blind, single-site behavioral intervention trial of adult patients with a diagnosis of bipolar disorder receiving care in the VA Ann Arbor Healthcare System. Up to 300 subjects will be enrolled, of which 150 will be randomized to receive the intervention and 150 will receive usual VA care. All subjects will complete a baseline clinical assessment and then subsequent follow-up assessments at 3, 6, 12, and 24 months. The intervention's three core components will be implemented by a nurse Care Manager and include: 1) self-management behavioral sessions for patients addressing the reduction of CVD risk factors through symptom control and behavior change based on Social Cognitive Theory, 2) care management to promote patient behavior change and coordinate care, and 3) implementation of practice guidelines for providers on management of CVD risk factors in patients with bipolar disorder. Medical and psychiatric care, including medications, will continue to be provided by the patient's usual providers. Usual VA care will be enhanced and consist of guideline implementation and general patient education (attention control), but will not include self-management sessions or Care Manager contacts. Primary clinical outcomes include changes in cholesterol, and health-related quality of life (SF-12 physical health summary score). Linear regression models will be used to determine the effect of the intervention on each outcome. Mediators of treatment effect including symptoms and health behaviors will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of bipolar disorder (I, II, not otherwise specified, or schizoaffective-bipolar subtype)
* Have a diagnosis or be at risk for arteriosclerotic cardiovascular disease (ASCVD).

We define this as a patient having a current diagnosis of or receiving treatment for at least one of the following medical conditions:

* hyperlipidemia or dyslipidemia (documented diagnosis or low-density lipoprotein >=160, or receiving statin or other treatment)
* hypertension (documented diagnosis or blood pressure of >=140/90 on 2 occasions)
* diabetes mellitus (documented diagnosis or HbA1C >=7%, or receiving treatment)
* obesity (documented diagnosis or BMI >30), based on medical record review of current problems
* current ASCVD diagnosis

Exclusion Criteria:

* Have unresolved substance intoxication or withdrawal, such as appearing to be intoxicated (e.g., incoherent, slurred speech), or experiencing withdrawal symptoms from substance abuse at the time of enrollment.
* Are already enrolled in a mental health program with a mobile outreach component in which clinical caregivers deliver services to the patient in the community (e.g., assertive community treatment or intensive case management). These patients may be receiving similar services to those offered in the intervention.
* Are unwilling or unable to provide informed consent or comply with study requirements at the time of enrollment (e.g., unable to complete forms or attend scheduled sessions due to serious illness or substantial functional limitations).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2008-05; Primary Completion 2012-05 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amy M. Kilbourne, PhD MPH, Principal Investigator — VA Ann Arbor Healthcare System
Locations (1):
- VA Ann Arbor Healthcare System, Ann Arbor, Michigan, United States

REFERENCES:
- [Derived] Kilbourne AM, Goodrich DE, Lai Z, Post EP, Schumacher K, Nord KM, Bramlet M, Chermack S, Bialy D, Bauer MS. Randomized controlled trial to assess reduction of cardiovascular disease risk in patients with bipolar disorder: the Self-Management Addressing Heart Risk Trial (SMAHRT). J Clin Psychiatry. 2013 Jul;74(7):e655-62. doi: 10.4088/JCP.12m08082. PMID 23945460

RESULTS

PARTICIPANT FLOW:
Groups:
- Chronic Care Model for Bipolar Disorder: An intervention group of patients with bipolar disorder and 1 or more risk factor for cardiovascular disease; group will receive self-management group sessions, followed by phone contacts by the Care Manager.
  Chronic care model involving self-management educational sessions, care management for up to 1 year, and guideline dissemination: The behavioral intervention is based on the Chronic Care Model (CCM) where patients receive information on managing bipolar symptoms and health habits in a group self-management session (up to 6 weekly sessions). The Care Manager then follows up with patients via phone contacts for 12 months following the intervention. The providers receive information on guidelines for care.
Period: Overall Study
Arm/Group | Chronic Care Model for Bipolar Disorder | Enhanced Usual Care
Started | 58 | 60
Completed | 35 | 40
Not Completed | 23 | 20

BASELINE CHARACTERISTICS:
Groups:
- Chronic Care Model for Bipolar Disorder: An intervention group of patients with bipolar disorder and 1 or more risk factor for cardiovascular disease (CVD); group will receive self-management group sessions, followed by phone contacts by the Care Manager.
  Chronic care model involving self-management educational sessions, care management for up to 1 year, and guideline dissemination: The behavioral intervention is based on the Chronic Care Model (CCM) where patients receive information on managing bipolar symptoms and health habits in a group self-management session (up to 6 weekly sessions). The Care Manager then follows up with patients via phone contacts for 12 months following the intervention. The providers receive information on guidelines for care.
- Enhanced Usual Care: A group of patients with bipolar disorder and one or more risk factors for cardiovascular disease (CVD) will be randomized to receive enhanced usual care. This group will receive usual care, plus mailings on wellness topics (attention control), and their providers will receive information on guideline concordant care.
- Total: Total of all reporting groups
Arm/Group | Chronic Care Model for Bipolar Disorder | Enhanced Usual Care | Total
Number analyzed (Participants) | 58 | 60 | 118
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.1 (10.6) | 52.4 (9.2) | 52.8 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 10 | 20
  Male | 48 | 50 | 98
Region of Enrollment [Number; unit: participants]
  United States | 58 | 60 | 118

OUTCOME MEASURES:

1. Primary Outcome: Systolic and Diastolic Blood Pressure (SBP, DBP)
Description: 24-month systolic and diastolic blood pressure (mm/Hg): lower is better
Time Frame: 24 months
Measure: Mean (Standard Deviation); unit: mm/Hg
Arm/Group | Chronic Care Model for Bipolar Disorder | Enhanced Usual Care
Number analyzed (Participants) | 58 | 60
mm/Hg
  24-month SBP in mm/Hg | 127.2 (15.4) | 130.4 (13.6)
  24-month DBP in mm/Hg | 75.9 (10.4) | 78.5 (10.3)
Statistical Analysis 1: Comparison: Chronic Care Model for Bipolar Disorder vs Enhanced Usual Care; Test type: Superiority or Other; p < .05, Mixed Models Analysis

2. Secondary Outcome: Manic Symptoms
Description: Manic symptoms based on the Internal State Scale (range is 0-500; higher score indicates more severe symptoms)
Time Frame: 24 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Chronic Care Model for Bipolar Disorder | Enhanced Usual Care
Number analyzed (Participants) | 58 | 60
units on a scale | 148.9 (120.9) | 173.4 (105.8)

3. Primary Outcome: Total Cholesterol
Description: Total cholesterol in mg/dl- lower is better
Time Frame: 24 months
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Chronic Care Model for Bipolar Disorder | Enhanced Usual Care
Number analyzed (Participants) | 58 | 60
mg/dL | 178.9 (45.5) | 175.9 (42.4)

4. Primary Outcome: Physical Health-related Quality of Life Score
Description: Physical health-related quality of life is based on the Short Form (SF)-12 survey physical health component (PCS) score- which ranges from 0 to 50, with higher scores indicating higher quality of life
Time Frame: 24 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Chronic Care Model for Bipolar Disorder | Enhanced Usual Care
Number analyzed (Participants) | 58 | 60
units on a scale | 36.8 (6.6) | 35.3 (7.0)

5. Secondary Outcome: Depressive Symptom Score
Description: Depressive symptoms based on the Internal State Scale (Range: 0-200, higher score = more severe symptoms)
Time Frame: 24 months
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Chonic Care Model for Bipolar Disorder: An intervention group of patients with bipolar disorder and 1 or more risk factor for cardiovascular disease; group will receive self-management group sessions, followed by phone contacts by the Care Manager.
  Chronic care model involving self-management educational sessions, care management for up to 1 year, and guideline dissemination: The behavioral intervention is based on the Chronic Care Model (CCM) where patients receive information on managing bipolar symptoms and health habits in a group self-management session (up to 6 weekly sessions). The Care Manager then follows up with patients via phone contacts for 12 months following the intervention. The providers receive information on guidelines for care.
Arm/Group | Chonic Care Model for Bipolar Disorder | Enhanced Usual Care
Number analyzed (Participants) | 58 | 60
units on a scale | 50.6 (46.4) | 60.3 (55.9)

6. Secondary Outcome: Disability Based on WHO-DAS Score
Description: Disability based on the WHO Disability Assessment Scale (WHO-DAS); range = 0-24, higher score equals greater disability
Time Frame: 24 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Chonic Care Model for Bipolar Disorder | Enhanced Usual Care
Number analyzed (Participants) | 58 | 60
units on a scale | 15.0 (10.9) | 16.5 (10.7)

7. Secondary Outcome: Body Mass Index (BMI)
Description: Body mass index (BMI) is reported in kilograms divided by meters squared (kg/m^2) with a normal (healthy) range of 18-24, in which >=25 is considered overweight, and >=30 is the definition of obesity
Time Frame: 24 months
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Chronic Care Model for Bipolar Disorder | Enhanced Usual Care
Number analyzed (Participants) | 58 | 60
kg/m^2 | 31.3 (5.8) | 33.4 (6.1)

ADVERSE EVENTS:
Groups:
- Arm 1: An intervention group of patients with bipolar disorder and 1 or more risk factor for cardiovascular disease; group will receive self-management group sessions, followed by phone contacts by the Care Manager.
  Chronic care model involving self-management educational sessions, care management for up to 1 year, and guideline dissemination: The behavioral intervention is based on the Chronic Care Model (CCM) where patients receive information on managing bipolar symptoms and health habits in a group self-management session (up to 6 weekly sessions). The Care Manager then follows up with patients via phone contacts for 12 months following the intervention. The providers receive information on guidelines for care.
- Arm 2: A group of patients with bipolar disorder and one or more risk factors for cardiovascular disease will be randomized to receive enhanced usual care. This group will receive usual care, plus mailings on wellness topics (attention control), and their providers will receive information on guideline concordant care.
Arm/Group | Arm 1 | Arm 2
Serious Adverse Events (participants affected / at risk) | 0/58 | 0/60
Other Adverse Events (participants affected / at risk) | 0/58 | 0/60

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes